CLINICAL TRIAL: NCT05426798
Title: Phase I Clinical Study of TQB2618 Injection in Combination With Demethylation Drugs in Patients With Recurrent/Refractory Acute Myeloid Leukemia, Myelodysplastic Syndromes
Brief Title: Clinical Study of TQB2618 Injection in Combination With Demethylation Drugs in Patients With Recurrent/Refractory Acute Myeloid Leukemia, Myelodysplastic Syndromes
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2618- I -02
Record Dates: First submitted 2022-06-16; First posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Recurrent/Refractory Acute Myeloid Leukemia, Myelodysplastic Syndromes
MeSH Terms: conditions — Recurrence; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Decitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2618 injection (Experimental): TQB2618 injection combined with demethylation drugs, 28 days as a treatment cycle until the disease progresses or the investigator judges that it is not suitable for subject to continue to take medicine.
  Interventions: Drug: TQB2618 injection azacitidine, AZA decitabine, DAC

INTERVENTIONS:
Drug: TQB2618 injection azacitidine, AZA decitabine, DAC — Drug1: TQB2618 injection is a novel tim-3 inhibitor.
  Drug2: Azacitidine (5-azacytidine) is a cytidine nucleoside analogue that selectively inhibits DeoxyriboNucleic Acid methyltransferases at low doses, resulting in gene promoter hypomethylation.
  Drug3: Decitabine is a cytidine deoxy nucleoside analogue that selectively inhibits DNA methyltransferases at low doses, resulting in gene promoter hypomethylation.

SUMMARY:
This project is an open, dose escalation and expansion phase I clinical study. The first phase is a dose escalation study, and the second phase is a dose expansion study based on the Maximum tolerated dose (MTD) / Recommended Phase II Dose (RP2D) obtained in the first phase. The purpose is to evaluate the tolerability and initially evaluate the antitumor efficacy of TQB2618 injection combined with demethylation drugs in patients with recurrent/refractory acute myeloid leukemia, myelodysplastic syndromes.

ELIGIBILITY:
Inclusion Criteria:

* 1 Subjects with medium-high risk recurrent/refractory International Prognostic Scoring System (IPSS-R) myelodysplastic syndromes(MDS) and acute myelocytic leukemia(AML) clearly diagnosed by pathology, who were intolerant to other medications and judged by the investigator to have no other appropriate treatment.
* 2 ≥18 years old; Eastern Cooperative Oncology Group (ECOG) physical status: 0-2; at least 3 months expected survival period.
* 3 The function of main organs is normal.
* 4 Subjects must need to adopt effective methods of contraception.
* 5 Subjects voluntarily joined the study, signed informed consent form, and with good compliance.

Exclusion Criteria:

* 1 Patients has had or is currently having other malignant tumors within 3 years. The following two conditions can be included in the group: other malignant tumors treated with a single operation to achieved 5 consecutive years of disease free survival (DFS)s. Cured cervical carcinoma in situ, non-melanoma skin cancer, nasopharyngeal carcinoma and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor infiltrating basement membrane)].
* 2 Patients diagnosed with acute promyelocytic leukemia or Philadelphia Chromosome-Positive Acute Myeloid Leukemia (Ph+AML) , or low-risk relapsed and refractory AML who only received second-line therapy;
* 3 The non-hematologic toxicity of previous antitumor treatment is not recovered to ≤ grade 1 (excluding hair loss).
* 4 Received major surgical treatment, open biopsy or obvious traumatic injury within 4 weeks before treatment.
* 5 The subjects had any history of bleeding or coagulopathy or who were being treated with anticoagulant.
* 6 Subjects had an arteriovenous thrombosis event within 6 months.
* 7 History of drug abuse, alcohol or drug abuse or mental disorder. Subjects who have epilepsy and require treatment.
* 8 Poor blood pressure control (systolic blood pressure ≥150mmHg or diastolic blood pressure ≥100 mmHg);
* 9 Subjects who had received allogeneic stem cell transplantation or autologous stem cell transplantation within 3 months；
* 10 Subjects with ≥ grade 2 myocardial ischemia or infarction, arrhythmia, prolonged QTc interval (including male QTc ≥450ms, female QTc ≥470ms) and ≥ grade 2 congestive heart failure with New York Heart Association (NYHA )classification；
* 11 Active or uncontrolled severe infection ≥common terminology criteria for adverse events （CTCAE） grade 2 infection)；
* 12 Subjects with active hepatitis.
* 13 The subjects was diagnosed with renal failure and required hemodialysis or peritoneal dialysis.
* 14 History of immunodeficiency, including positive human immunodeficiency virus (HIV) test or other acquired, congenital immunodeficiency disease, or history of organ transplantation.
* 15 Poor control of diabetes (fasting glucose GLU > 10mmol/L);
* 16 Subjects who have received radiation therapy or the treatment of proprietary Chinese medicines with anti-tumor indications clearly stated in the National Medical Products Administration (NMPA) approved drug instructions within 4 weeks of starting treatment.
* 17 Uncontrolled pleural effusion, pericardial effusion or ascites;
* 18 Subjects with central nervous system aggression;
* 19 Vaccination history of live attenuated vaccine before 4 weeks of starting treatment, or planned vaccination of live attenuated vaccine during the study period.
* 20 History of severe allergy to study drugs and pharmaceutical excipients .
* 21 Subjects diagnosed with active autoimmune disease within 2 years before starting treatment.
* 22 Receiving any other investigational agent within 4 weeks before first dose.
* 23 According to the investigator's judgment, there are concomitant diseases that seriously endanger the safety of the subject or affect the completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2022-04-29 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Baseline up to 78 weeks
  To evaluate MTD of TQB2618 injection combined with demethylation drugs in patients with recurrent/refractory acute myeloid leukemia, myelodysplastic syndromes.
Dose limited toxicity (DLT) | Baseline up to 78 weeks
  To evaluate DLT of TQB2618 injection combined with demethylation drugs in patients with recurrent/refractory acute myeloid leukemia, myelodysplastic syndromes.
Recommended Phase II Dose (RP2D) | Baseline up to 78 weeks
  To evaluate RP2D of TQB2618 injection combined with demethylation drugs in patients with recurrent/refractory acute myeloid leukemia, myelodysplastic syndromes.
Objective Response Rate | Baseline up to 78 weeks
  To evaluate ORR of TQB2618 injection combined with demethylation drugs in patients with recurrent/refractory acute myeloid leukemia, myelodysplastic syndromes.

SECONDARY OUTCOMES:
Adverse events (AE) | Baseline up to 92 weeks
  incidence and severity of adverse events (AE)
Receptor occupation (RO) | Baseline up to 92 weeks
  Receptor occupation (RO) of Tim-3 after administration
anti-drug antibody (ADA)/ neutralizing antibody (Nab) | Baseline up to 92 weeks
  Immunogenicity related indicators: the incidence and titer of the subjects' anti-drug antibody (ADA) and the incidence of neutralizing antibody (Nab);
Progress Free Survival (PFS) Progress Free Survival (PFS) | up to 92weeks
  Time from the first dose to the first documentation of progressive disease (PD) or death from any cause, whichever occurs first
Disease control rate (DCR) | up to 92weeks
  Percentage of participants achieving complete response (CR) and partial response (PR) and stable disease (SD).
Duration of Response (DOR) | up to 92weeks
  The time when the participants first achieved complete or partial remission to disease progression.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China